CLINICAL TRIAL: NCT01117415
Title: Cost Effectiveness Analysis of Transgastric Cholecystectomy, Transvaginal Cholecystectomy, and Laparoscopic Cholecystectomy: Projected Long Term Outcomes and Complications Evaluation
Brief Title: Cost Effectiveness Analysis of Cholecystectomy, Projected Long Term Outcomes and Complications Evaluation
Acronym: NOTES
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Marks, MD, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: 09-07-40; 09-07-40 (Other: University Hospital case Medical Center)
Record Dates: First submitted 2010-04-12; First posted 2010-05-05 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Cholelithiasis
Keywords: Gall Bladder; Cholecystectomy
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gall Bladder Surgery: Who have symptomatic cholelithiasis and wish to undergo laparoscopic cholecystectomy for treatment.

SUMMARY:
Participation in this research study does not involve any procedures. Health preference will be ascertained through standard techniques including time-tradeoff, standard gamble, and rating scale to assess risks regarding potential complications specific to NOTES (Natural Orifice Translumenal Endoscopic Surgery)gallbladder removal.

DETAILED DESCRIPTION:
The enticement of scarless surgery has created an unprecedented wave of enthusiasm and collaboration amongst surgeons, gastroenterologists, industry, and the lay public. However, major hurdles remain between current minimally invasive practices and the ultimate goal of safe, effective Natural Orifice Translumenal Endoscopic Surgery (NOTES). In an ideal world, these procedures should incur equivalent (or less) morbidity than current laparoscopic approaches and offer benefits of incisionless surgery. This idealism has been quickly tempered by the potential to create new and devastating complications with only minimal potential benefit to the patient. Several critical questions need to be answered. What probability of complication(s) are to be accepted? How will the potential benefits of NOTES be weighed against these new complications? What factors unique to NOTES will contribute to its cost effectiveness? The proposed study seeks to answer these questions before they occur. These results will give clinicians and investigators the necessary information with which to compare outcomes of NOTES and potentially alter techniques for safer, more effective interventions.

ELIGIBILITY:
Inclusion Criteria:

* Candidate of either sex
* 18 years old or above
* Have symptomatic cholelithiasis
* Wish to undergo laparoscopic cholecystectomy for treatment

Exclusion Criteria:

* Not Applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the University Hospitals Case Medical Center Department of Surgery. The patient population in this study for the visual analog scale measurement, standard gamble questionnaire, and time trade-off questionnaire will be candidates of either sex, 18 years old or above, who have symptomatic cholelithiasis and wish to undergo laparoscopic cholecystectomy for treatment. The patients will be asked to participate in the study after evaluation by either the principal investigator, co-investigators, or study coordinator. The investigator will discuss the study with the patient and the study coordinator will participate in reviewing details and questions regarding the study if necessary. Patients will be recruited until 40 participants are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2007-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Compare cost effectiveness data at one year postoperative | 1 year
  One year cost effectiveness data comparing transgastric cholecystectomy, transvaginal cholecystectomy, and laparoscopic cholecystectomy. Costs from two national databases: the State Ambulatory Surgery Database (SASD) and the NIS. The main outcome measure for this study will be cost per quality adjusted life year (QALY). Markov modeling techniques for model patient experiences for each of the procedures analyzed. Monte Carlo simulation will be used to calculate cost per QALY over a one year time span with determination of the incremental cost effectiveness ratio.

SECONDARY OUTCOMES:
Analyze the important factor that contributes to cost effectiveness at one year post operative. | One year
  Extensive sensitivity analyses of how individual factors (e.g. probability of gastric leak in transgastric cholecystectomy) impact cost effectiveness. Factors are varied over a clinically plausible range and their impact on cost effectiveness determined. One way and two way sensitivity analyses allow alterations of one or two factors simultaneously. Multiway sensitivity analysis using Monte Carlo simulation will be used to vary several variables simultaneously and to determine impact on cost effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin K. Poulose, MD, MPH, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States